CLINICAL TRIAL: NCT05821985
Title: Evaluation of the Effect of Dextrose Prolotherapy Versus Dry Needling Therapy for the Treatment of Temporomandibular Joint Anterior Disc Displacement With Reduction (A Randomized Controlled Trial)
Brief Title: Evaluation of the Effect of Dextrose Prolotherapy Versus Dry Needling Therapy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Beni-Suef University (Other)
Responsible Party: Principal Investigator, Ahmed Nagi Alghandour, Lecturer, Beni-Suef University
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: 3
Record Dates: First submitted 2023-03-29; First posted 2023-04-20 (Actual); Last update posted 2024-05-03 (Actual); Status verified 2024-05

CONDITIONS: Temporomandibular Joint Disorders
MeSH Terms: conditions — Temporomandibular Joint Disorders

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- The Study group (Other): The patients within the study group will receive intraarticular TMJ and masseteric Trigger point injection of a solution that contains (0.75 ml. 12.5% Dextrose solution, 0.75 ml. Saline solution, and 1.5 ml. Lidocaine).
  Interventions: Procedure: The study group
- The Control group (Other): Patients in the control group will receive intraarticular TMJ and masseteric Trigger point dry needle insertion without injecting any solution.
  Interventions: Procedure: The Control group

INTERVENTIONS:
Procedure: The study group — The patients within the study group will receive intraarticular TMJ and masseteric Trigger point injection of a solution that contains (0.75 ml. 12.5% Dextrose solution, 0.75 ml. Saline solution, and 1.5 ml. Lidocaine). Each patient will receive four injections at two-week intervals, aided by a 25 gauge needle connected to a 3 ml. plastic syringe.
  Arms: The Study group
Procedure: The Control group — The Control group:
  Patients in the control group will receive intraarticular TMJ and masseteric Trigger point dry needle insertion without injecting any solution. Each patient will receive four dry needle insertions at two-week intervals, aided by a 25-gauge and 3.8 cm length needle.
  i.e., All the patients will be subjected to intraarticular needle insertion. However, only the patients within the study group will be injected with the Dextrose Prolotherapy solution.
  Arms: The Control group

SUMMARY:
The hypertonic dextrose injection; Prolotherapy is a proliferation injection therapy that aims to trigger a low-grade inflammatory response inside the (TMJ), with the resultant captivation of abundant fibroblasts that regenerate and strengthen the tendinous and ligamentous attachments and stabilize the disc and the fibro-osseous junctions.

On the other hand, dry needling' refers to the insertion of needles without the use of injectate. Dry needling is beneficial for treating a variety of neuromusculoskeletal pain syndromes as it represents a treatment modality for the ligaments and tendons, muscles, subcutaneous fascia, peripheral nerves, and neurovascular bundles. Deep dry needling (DDN) is a technique that utilizes the Intracapsular insertion of dry needles to approach the discal insertion to the lateral pterygoid muscle and the masseteric muscle origin, along the zygomatic bone and arch, aiming to inactivate the muscular trigger points (TPs).

DETAILED DESCRIPTION:
The Temporomandibular joint (TMJ) represents the most complex synovial articulation in the human body, with its articular disc enclosed between the articular tubercle's slope and the convexity of the mandibular condyle.

Although the Magnetic resonance interpretation of the normal discal position defines the posterior discal band atop the highest convexity of the mandibular condyle, at a 12 o'clock position, this discal disposal is altered in almost 30% of the population without physical signs. Which rendered the treatment of the discal displacement mainly dependent on alleviating the signs and symptoms rather than restoring the anatomical disc position.

Various non-invasive therapeutic modalities are utilized for relieving the signs and symptoms of anterior discal displacement, including physical therapy, exercises, ischemic compression, heat therapy, acupuncture, dry needling, wet needling injections with different agents, and pharmacological treatments.

Among those, the trigger point injection is an effective modality, with or without the injection of saline or ringer's solutions, hyaluronic acid, corticosteroids, local anesthetics, botulinum toxin, platelet-rich plasma, or hypertonic dextrose The current study aims to design a randomized controlled trial that compares the effect of injecting 12.5 % of dextrose solution intraarticular and into the myofascial trigger points versus the dry needling of the same sites on alleviating the clinical signs and symptoms of (TMJ) disc displacement with reduction.

ELIGIBILITY:
Inclusion Criteria:

1. Patients of both genders with an age group of 18-45 years.
2. Those patients with the radiographic interpretation of temporomandibular joint disc displacement with reduction (MRI) and the clinical signs of pain, limitation of mouth opening, and TMJ clicking.
3. The presence of associated myofascial pain with masseteric trigger points (TPs)

Exclusion Criteria:

1. Any previous temporomandibular joint treatment.
2. Any systemic disease affecting the temporomandibular joint's anatomy, mechanical function, or outcome of the proposed treatment.
3. Those Patients with a history of allergic reactions to any components of the injectable solution

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2023-09-01 (Actual); Primary Completion 2024-03-01 (Actual); Study Completion 2024-04-01 (Actual)

PRIMARY OUTCOMES:
Pain threshold | 8 months
  by using visual analogue scale from 0 to 10 which 10 is the worst pain
Interincisal opening | 8 months
  distance by cm caliber from the between the anterior teeth at the maximal unassisted nonpainful opening of the patient.
clicking | 8 months
  (evident or not)

CONTACTS AND LOCATIONS:
Locations (1):
- Beni-suef university, Banī Suwayf, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Gibaly A, Abdelmoiz M, Alghandour AN. Evaluation of the effect of dextrose prolotherapy versus deep dry needling therapy for the treatment of temporomandibular joint anterior disc displacement with reduction: (a randomized controlled trial). Clin Oral Investig. 2024 Aug 8;28(9):475. doi: 10.1007/s00784-024-05830-z. PMID 39115583